CLINICAL TRIAL: NCT01415869
Title: Occult Gastrointestinal Bleeding in Non-pulsatile Left Ventricular Assist Device(VAD)Patients
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joseph L. Blackshear, PI, Mayo Clinic
Other Study IDs: 11-003334
Record Dates: First submitted 2011-08-01; First posted 2011-08-12 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Gastrointestinal Bleeding; Complication of Internal Device
Keywords: Ventricular Assist Device; Gastrointestinal Bleeding; VAD
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cross Sectional: Patients with implanted non-pulsatile ventricular assist devices of any type and at any time after implantation
- Prospective: Patients with usual VAD indications will be invited to participate, when, in the opinion of their treating physician a VAD will be highly likely within one month.

SUMMARY:
The purpose of this study is to estimate the proportion of Ventricular Assist Device (VAD) patients with abnormal gastrointestinal bleeding as assessed by HemoQuant fecal occult blood test. Also, in patients with gastrointestinal bleeding present, to summarize the extent of gastrointestinal bleeding; to examine the behavior of HemoQuant fecal occult blood test over time by estimating the proportion of VAD patients with a positive test prior to implantation; at one week, one month, three months, six months and one year post implantation, and after explantation of the VAD and to evaluate whether presence of any abnormal fecal HemoQuant test is predictive of a future major bleeding event.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 - cross sectional study. Patients with implanted non-pulsatile ventricular assist devices of any type and at any time after implantation
* Group 2 - prospective study. Patients with usual VAD indications will be invited to participate, when, in the opinion of their treating physician a VAD will be highly likely within one month.

Exclusion Criteria:

* Unwillingness to provide stool samples for study
* Unwillingness to be followed for study endpoints.
* Unwillingness to follow dietary restrictions necessary for accurate HemaQuant measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Group 1 Patients with implanted non-pulsatile ventricular assist devices of any type and at any time after implantation
  * Group 2 Patients with usual VAD indications will be invited to participate, when, in the opinion of their treating physician a VAD will be highly likely within one month.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2011-06-22 (Actual); Primary Completion 2013-06-22 (Actual); Study Completion 2013-06-22 (Actual)

PRIMARY OUTCOMES:
Proportion of VAD Patients with Gastrointestinal Bleeding as Assessed by HemoQuant Fecal Occult Blood Testing | 1 year
  We will estimate the proportion of VAD patients with gastrointestinal bleeding as assessed by HemoQuant fecal occult blood test along with an exact binomial 95% confidence interval (CI). HemoQuant values will be summarized using the sample median, minimum, 25th percentile, 75th percentile, and maximum. These measures will be reported overall, regardless of time after implantation, in order to provide an estimate of the frequency of gastrointestinal bleeding in VAD patients that will be able to be published quickly and raise awareness of this issue.

SECONDARY OUTCOMES:
Examine Behavior of Gastrointestinal Bleeding in VAD Patients By Estimating the Proportion of VAD Patients with an Abnormal HemoQuant Test Prior to Implantation | 1 year
  We will examine the behavior of gastrointestinal bleeding over time in VAD patients (as assessed by HemoQuant fecal occult blood test), by estimating the proportion of VAD patients with an abnormal HemoQuant test (and 95% CI) prior to implantation; at one week, one month, three months, six months and one year post implantation, and after explantation of the VAD.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Blackshear, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials